CLINICAL TRIAL: NCT06749678
Title: Effect of Prehabilitation During the Conversion Therapy on Postoperative Outcomes in Patients With Unresectable Hepatocellular Carcinoma: a Prospective, Open, Randomized Controlled Trial
Brief Title: Effect of Prehabilitation During the Conversion Therapy on Postoperative Outcomes in Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-994-03
Record Dates: First submitted 2024-12-05; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC); Prehabilitation
Keywords: unresectable hepatocellular carcinoma; prehabilitation; conversion therapy
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): In addition to routine nursing measures, the prehabilitation group underwent prehabilitation measures during the conversion therapy period.
  Interventions: Behavioral: Prehabilitation; Behavioral: Routine nursing measures
- Control group (Placebo Comparator): During the conversion therapy period, the control group only took routine nursing measures.
  Interventions: Behavioral: Routine nursing measures

INTERVENTIONS:
Behavioral: Prehabilitation — In addition to routine nursing measures, the prehabilitation group underwent prehabilitation measures during the conversion therapy period. It includes the following strategies: (1) Exercise: Exercise should be carried out when the patient's condition allows, and the exercise programme should be dynamically adjusted according to the patient's tolerance, and it is advisable to maintain the Borg score between 11~13 points (i.e., subjectively feel relaxed or a little strained). (2) Nutritional support: ensure that the patient's daily energy intake is 20~25kcal/kg (the target energy reaches 30~35kcal/kg), and the protein intake is 1.2~1.5g/(kg·d). (3) Psychological intervention: for patients with mild to moderate anxiety or depression, health education, music therapy and other psychological interventions are carried out. For patients with severe anxiety or depression, psychologists will conduct psychological consultation for patients and provide professional psychological therapy.
  Arms: Prehabilitation group
Behavioral: Routine nursing measures — Routine nursing measures including: (1) general education: for different patients, cards and manuals were used to focus on the diagnosis and treatment matters such as examination, treatment, surgery and perioperative treatment, so as to alleviate the anxiety and fear of patients and better cooperate with hospital management. (2) Medical optimization: including smoking cessation, alcohol restriction, chronic disease control, etc. (3) Nutritional support: Routine dietary guidance and nutritional support are given, and intravenous or oral nutrition therapy is given to patients who are emaciated and have lost more than 3kg in the past one month. (4) Rehabilitation training: Carry out rehabilitation training education and guidance, including fist exercises, chest expansion exercises, deep breathing, sputum discharge, abdominal muscle strengthening training, etc.

SUMMARY:
This is a prospective, randomised controlled clinical trial to study the impact of prehabilitation on postoperative complications, physical function, quality of life, and short-term survival outcomes in patients with unresectable liver cancer undergoing conversion therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be aged between 18 and 75 years, inclusive, with no gender restrictions.
2. Patients must have an initial diagnosis of unresectable hepatocellular carcinoma (HCC) confirmed by EASL/AASLD diagnostic criteria, pathological histology, or cytology, and must be planned for conversion therapy.
3. Patients must have an American Society of Anesthesiologists (ASA) physical status classification of ≤III.
4. Patients must be physically capable of participating in exercise training, defined as the ability to walk continuously on flat ground for more than 200 meters without rest and to climb two flights of stairs consecutively without requiring a break.
5. Patients must not have any psychiatric disorders, speech impediments, or consciousness disturbances, and must possess adequate comprehension, communication, and literacy skills.
6. Patients must voluntarily enroll in the study, be able to provide written informed consent, and be capable of understanding and adhering to the trial protocol and follow-up procedures.

   -

Exclusion Criteria:

1. A known diagnosis of cholangiocarcinoma, sarcomatoid hepatocellular carcinoma (HCC), combined hepatocellular carcinoma, or fibrolamellar carcinoma.
2. Presence of extrahepatic metastases or concurrent other malignant tumors.
3. Presence of psychiatric disorders or cognitive impairments that would impede compliance with study requirements.
4. Unsuitability for participation in exercise training due to skeletal muscle diseases or a history of fracture within the past 6 months.
5. Pregnant or breastfeeding women.
6. Individuals with severe and irreversible cardiac, pulmonary, or renal organic diseases, or severe anemia, which would make them unsuitable for preoperative rehabilitation programs. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Complication Composite Index (CCI) at 30 days postoperatively | 30 days after surgery
  Surgical patients were scored based on the severity and number of complications that occurred within 30 days after surgery.

SECONDARY OUTCOMES:
30-Day Postoperative Mortality Rate | 30 days after surgery
  The 30-day postoperative mortality rate refers to the proportion of patients who die within 30 days following surgery. This rate was recorded separately for patients in both groups who underwent the surgical procedure.
Six-Minute Walk Distance (6MWD) | Baseline, each cycle of therapy, the time of surgery, and at 2、6 weeks and 6 months postoperatively.
  In a flat, straight corridor, a 6-minute walk test is conducted to measure the total distance covered on foot.
The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | Baseline, each cycle of therapy, the time of surgery, and at 2、6 weeks and 6 months postoperatively
  The EORTC QLQ-C30 questionnaire, comprising 30 items, is meticulously structured into multiple dimensions or domains to provide a comprehensive evaluation of the quality of life in cancer patients. Patients respond to each item based on their personal circumstances, with each item assigned a specific scoring range, typically from 0 to 4 points (or 0 to 3 points, depending on the particular configuration of the item).
The Generalized Anxiety Disorder 7-item scale (GAD-7) Score | Baseline, each cycle of therapy, the time of surgery, and at 2、6 weeks and 6 months postoperatively
  The Generalized Anxiety Disorder-7 (GAD-7) scale consists of seven items, each of which is associated with symptoms of anxiety. These items include feelings of being nervous, anxious, or on edge; not being able to stop or control worrying; worrying too much about various things; finding it hard to relax; being restless due to unease; becoming easily annoyed or irritable; and feeling afraid as if something awful might happen. Patients respond to each item based on their personal circumstances.
The Patient Health Questionnaire-9 (PHQ-9) Depression Scale Score | Baseline, each cycle of therapy, the time of surgery, and at 2、6 weeks and 6 months postoperatively
  The Patient Health Questionnaire-9 (PHQ-9) comprises nine items, each addressing a distinct facet of depressive symptoms. The total score is derived by aggregating the scores from each individual item based on the respondent's chosen answers.
The incidence and severity of postoperative complications. | 30 days after surgery
  During the course of this study and throughout the follow-up period, the severity of postoperative complications in patients who underwent surgery in both groups will be graded and assessed according to the Clavien-Dindo classification system, with all occurrences and degrees of severity of complications being documented.
Adverse Events Related to Conversion Therapy | Up to approximately 2 years
  During the course of this study and throughout the follow-up period, the severity of adverse events will be graded and assessed according to the NCI-CTCAE 5.0. All occurrences of adverse events (AEs), treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs) will be documented, including their incidence, severity, and correlation with the study medication. Additionally, the number and proportion of subjects who discontinue treatment due to these adverse events will be recorded.
Objective Response Rate (ORR) | Up to approximately 2 years
  Objective Response Rate (ORR) is a term used in oncology to describe the proportion of patients who experience a complete or partial reduction in their tumor burden in response to treatment. This measure includes both complete responses (CR) and partial responses (PR), and is an important endpoint in assessing the efficacy of cancer therapies.
Progression-Free Survival (PFS) | Up to approximately 2 years
  The time from the initiation of the conversion treatment protocol to the occurrence of tumor progression (in any aspect) or death (for any reason).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No